CLINICAL TRIAL: NCT01416688
Title: S1013: A Prospective Study of Epidermal Growth Factor Receptor (HER-1/EGFR) Inhibitor-Induced Dermatologic Toxicity: Validation of the Functional Assessment of Cancer Therapy-EGFRI 18(FACT-EGFRI 18) Questionnaire for EGFRI-Induced Skin Toxicities
Brief Title: S1013: Validation of Cancer Questionnaire for Skin Toxicities in Patients With Colorectal Cancer or Lung Cancer Receiving Cetuximab, Panitumumab, or Erlotinib Hydrochloride
Status: Completed | Type: Observational
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: S1013; S1013 (Other: SWOG); U10CA037429 (NIH); NCI-2011-02983 (Other: NCI)
Record Dates: First submitted 2011-08-12; First posted 2011-08-15 (Estimated); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Colorectal Cancer; Dermatologic Complications; Lung Cancer; Therapy-related Toxicity
Keywords: therapy-related toxicity; dermatologic complications; stage I colon cancer; stage IIA colon cancer; stage IIB colon cancer; stage IIC colon cancer; stage IIIA colon cancer; stage IIIB colon cancer; stage IIIC colon cancer; stage IVA colon cancer; stage IVB colon cancer; stage I rectal cancer; stage IIA rectal cancer; stage IIB rectal cancer; stage IIC rectal cancer; stage IIIA rectal cancer; stage IIIB rectal cancer; stage IIIC rectal cancer; stage IVA rectal cancer; stage IVB rectal cancer; stage IA non-small cell lung cancer; stage IB non-small cell lung cancer; stage IIA non-small cell lung cancer; stage IIB non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; extensive stage small cell lung cancer; limited stage small cell lung cancer; recurrent small cell lung cancer; recurrent colon cancer; recurrent rectal cancer; recurrent non-small cell lung cancer
MeSH Terms: conditions — Colorectal Neoplasms; Lung Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — Psychiatric Rehabilitation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Observation and Questionnaires: Patients will be given questionnaires for the assessment of therapy complications, psychosocial assessment and care, and quality-of-life assessment.
  Interventions: Procedure: assessment of therapy complications; Procedure: psychosocial assessment and care; Procedure: quality-of-life assessment

INTERVENTIONS:
Procedure: assessment of therapy complications — Will be given by questionnaire
Procedure: psychosocial assessment and care — Will be given by questionnaire
Procedure: quality-of-life assessment — Will be given by questionnaire

SUMMARY:
RATIONALE: Questionnaires that patients can use to assess skin toxicities related to treatment may help identify the intermediate-and long-term effects of cetuximab, panitumumab, or erlotinib hydrochloride.

PURPOSE: This trial studies the validation of a cancer questionnaire for skin toxicities in patients with colorectal or lung cancer receiving cetuximab, panitumumab, or erlotinib hydrochloride.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To establish psychometric properties for the Functional Assessment of Cancer Therapy Epidermal Growth Factor Receptor Inhibitor (FACT-EGFRI 18) module (based on criterion validity, known group's validity, internal consistency reliability, and responsiveness to change) as a patient-reported outcome (PRO) measure of EGFRI-induced skin-related toxicity.

Secondary

* To document minimally important differences over time for the FACT-EGFRI 18 by comparing mean changes in this PRO measure to the patient's direct assessment of change using two anchor items (change in skin condition severity and impact).
* To examine the association between toxicity profiles (severity and time to onset), and treatment profiles (e.g., delays and discontinuation) and the FACT-EGFRI 18 scores.
* To assess degree of concordance between FACT-EGFRI 18 ratings and study site physician CTCAE Version 4.0 EGFRI-Induced Dermatologic Toxicity Grading Assessment ratings.
* To evaluate feasibility outcomes.

OUTLINE: This is a multicenter study.

Patients complete the S1013 Functional Assessment of Cancer Therapy Epidermal Growth Factor Receptor Inhibitor (FACT-EGFRI 18) at baseline and prior to beginning therapy and clinical assessment. Patients also complete FACT-EGFRI 18 and the Changes in Skin Symptoms on days 1*, 8**, 15, 22, 29, 36, 43, 71, 99, and 127. Patients who do not develop any grade of papulopustular rash within 42 days are removed from study.

Investigators performing the patients' clinical assessment complete the EGFRI-Induced Dermatologic Toxicity Grading Assessment on days 1, 8, 15, 22, 29, 36, 43, 71, 99, and 127, and the Treatment Form assessment on days 22, 43, 71, 99, and 127. Nurses or clinical trial administrators (CRA) also complete the S1013 Cover Sheet for Patient Complete Questionnaires accompanying the FACT-EGFRI 18 patients' questionnaires at each schedule assessment.

NOTE: *Patients start EGFRI therapy.

NOTE: **Change in Skin Symptoms questionnaire starts on Day 8.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Patients must have a diagnosis of colorectal or lung cancer and be planning to receive one of the following epidermal growth factor receptor (HER1/EGFR) inhibitor therapies listed below for at least 6 weeks:

  * Cetuximab 400 mg/m² loading dose, 250 mg/m² weekly
  * Cetuximab 500 mg/m² every 2 weeks
  * Panitumumab 6 mg/kg every 2 weeks
  * Erlotinib hydrochloride 100-150 mg daily
  * Other HER1/EGFR inhibitor therapies, schedules, or doses of the above listed agents are not allowed
  * Concurrent chemotherapy and other anti-cancer therapies (such as carboplatin, paclitaxel, and bevacizumab) are allowed EXCEPT for the following chemotherapeutic agents that are known to cause skin rash that could interfere with EGFRI-induced skin toxicity assessment: gemcitabine, capecitabine, and topical fluorouracil (Efudex™, Fluoroplex™, Carac™)
* Patients must have completed the baseline S1013 Functional Assessment of Cancer Therapy- (FACT) EGFRI 18 within 7 days prior to registration

PATIENT CHARACTERISTICS:

* Patients must have a Zubrod performance status of 0-2
* Patients must not have any of the following serious concomitant skin disorders that, in the investigator's opinion, could interfere with assessment of epidermal growth factor receptor inhibitor (EGFRI)-induced skin toxicity: atopic dermatitis [eczema]; contact dermatitis; psoriasis; rosacea; severe photosensitivity; scleroderma; steroid-induced acne; or xerosis
* Patients must be able to complete questionnaires in English

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Patients may have had prior epidermal growth factor receptor (HER1/EGFR) inhibitor therapy but must have fully recovered from any skin toxicities prior to registration
* Patients must not be planning to receive any of the following concomitant medications that can cause skin rash or other dermatologic reactions that could interfere with the EGFRI-induced skin toxicity assessments, for the duration of the study: allopurinol; systemic corticosteroids; topical retinoids (Retin-A™, Tretinoin™); or oral retinoids (Amnesteem™, Claravis™, Sotret™)
* Patients must not be planning to receive concurrent external-beam radiation therapy, including prophylactic cranial radiation
* Patients may concurrently participate in other therapeutic clinical trials

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Limited institutions from the SWOG membership.
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2011-11-15 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2019-04-08 (Actual)

PRIMARY OUTCOMES:
Psychometric properties of the FACT-EGFRI 18 | 127 days from registration

SECONDARY OUTCOMES:
Change in severity and impact of skin symptoms | 127 days from registration
Agreement between site physician ratings with the CTCAE Version 4 and patient ratings for the FACT-EGFRI 18 items | 127 days from registration
Associations between toxicity profile and treatment profiles | 127 days from registration
Feasibility as measured by accrual, time to specified accrual, time to complete forms | 2 years from study activation

CONTACTS AND LOCATIONS:
Overall Officials: Laurence H. Baker, DO, FACOI, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (113):
- United States (113):
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - The University of Arizona Medical Center-University Campus, Tucson, Arizona
  - East Bay Radiation Oncology Center, Castro Valley, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Epic Care-Dublin, Dublin, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - El Camino Hospital, Mountain View, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Hematology and Oncology Associates-Oakland, Oakland, California
  - Doctors Medical Center- JC Robinson Regional Cancer Center, San Pablo, California
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Cancer Care Center of Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Little Company of Mary Hospital, Evergreen Park, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Cancer Care Specialists of Illinois-Swansea, Swansea, Illinois
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - University Health-Conway, Monroe, Louisiana
  - Louisiana State University Health Sciences Center Shreveport, Shreveport, Louisiana
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - Singh and Arora Hematology Oncology PC, Flint, Michigan
  - McLaren Cancer Institute-Lapeer Region, Lapeer, Michigan
  - McLaren Cancer Institute-Macomb, Mount Clemens, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Capital Region Medical Center-Goldschmidt Cancer Center, Jefferson City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Winthrop University Hospital, Mineola, New York
  - Columbia University/Herbert Irving Cancer Center, New York, New York
  - Cancer Care of Western North Carolina, Asheville, North Carolina
  - Mission Hospital-Memorial Campus, Asheville, North Carolina
  - Hope Women's Cancer Centers-Asheville, Asheville, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Carolinas HealthCare System NorthEast, Concord, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Hendersonville Hematology and Oncology at Pardee, Hendersonville, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - High Point Regional Hospital, High Point, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Carolinas HealthCare System Union, Monroe, North Carolina
  - Carolinas HealthCare System Cleveland, Shelby, North Carolina
  - Southeastern Medical Oncology Center-Wilson, Wilson, North Carolina
  - Southeast Clinical Oncology Research (SCOR) Consortium NCORP, Winston-Salem, North Carolina